CLINICAL TRIAL: NCT01134042
Title: HZA106829: A Randomised, Double-blind, Parallel Group, Multicentre Study of Fluticasone Furoate/GW642444 Inhalation Powder, Fluticasone Furoate Inhalation Powder Alone, and Fluticasone Propionate Alone in the Treatment of Persistent Asthma in Adults and Adolescents
Brief Title: Study HZA106829: Efficacy/Safety Study of Fluticasone Furoate/Vilanterol (GW642444) in Adult and Adolescent Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106829
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Fluticasone propionate; asthma; vilanterol; GW642444; Fluticasone furoate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone Furoate/Vilanterol (Experimental): Fluticasone furoate/vilanterol inhalation powder once daily + Placebo inhalation powder twice daily for 24 weeks
  Interventions: Drug: Fluticasone Furoate/Vilanterol Inhalation Powder; Other: Placebo Inhalation Powder 2
- Fluticasone Furoate (Active Comparator): Fluticasone furoate inhalation powder once daily + Placebo inhalation powder twice daily for 24 weeks
  Interventions: Drug: Fluticasone Furoate Inhalation Powder; Other: Placebo Inhalation Powder 2
- Fluticasone Propionate (Active Comparator): Fluticasone propionate inhalation powder twice daily + Placebo inhalation powder once daily for 24 weeks
  Interventions: Drug: Fluticasone Propionate Inhalation Powder; Other: Placebo Inhalation Powder 1

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol Inhalation Powder — Fluticasone furoate/Vilanterol inhalation powder inhaled orally once daily for 24 weeks
  Arms: Fluticasone Furoate/Vilanterol
Drug: Fluticasone Furoate Inhalation Powder — Fluticasone furoate inhalation powder inhaled orally once daily for 24 weeks
  Arms: Fluticasone Furoate
Drug: Fluticasone Propionate Inhalation Powder — Fluticasone propionate inhalation powder inhaled orally twice daily for 24 weeks
  Arms: Fluticasone Propionate
Other: Placebo Inhalation Powder 1 — Placebo in novel dry powder inhaler once daily
  Arms: Fluticasone Propionate
Other: Placebo Inhalation Powder 2 — Placebo in Diskus inhaler twice daily
  Arms: Fluticasone Furoate; Fluticasone Furoate/Vilanterol

SUMMARY:
The purpose of the study is to compare the efficacy and safety of fluticasone furoate/vilanterol (GW642444) inhalation powder administered once daily each evening with fluticasone furoate inhalation powder administered alone once daily each evening in adolescent and adult subjects 12 years of age and older with persistent bronchial asthma over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at least 12 years of age
* Both genders; females of childbearing potential must be willing to use birth control method
* Pre-bronchodilator FEV1 of 40-90% predicted
* Reversibility FEV1 of at least 12% and 200mls
* Current asthma therapy that includes an inhaled corticosteroid for at least 12 weeks prior to first visit

Exclusion Criteria:

* History of life-threatening asthma
* Respiratory infection or oral candidiasis
* Asthma exacerbation within 12 weeks
* Concurrent respiratory disease or other disease that would confound study participation or affect subject safety
* Allergies to study drugs, study drugs' excipients, medications related to study drugs
* Taking another investigational medication or medication prohibited for use during this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- United States (22):
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Sugar Land, Texas
- Germany (10):
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
- Japan (10):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Działdowo
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Piekary Śląskie
  - GSK Investigational Site, Sopot
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (7):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kosinski M, Nelsen L, Rizio AA, Lay-Flurrie J, von Maltzahn R, Jacques L, Schatz M, Stanford RH, Svedsater H. Psychometric properties of the Asthma Control Test in 2 randomized clinical trials. J Allergy Clin Immunol Pract. 2021 Jan;9(1):561-563.e1. doi: 10.1016/j.jaip.2020.07.040. Epub 2020 Aug 6. No abstract available. PMID 32771685
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Gross AS, Goldfrad C, Hozawa S, James MH, Clifton CS, Sugiyama Y, Jacques L. Ethnic sensitivity assessment of fluticasone furoate/vilanterol in East Asian asthma patients from randomized double-blind multicentre Phase IIb/III trials. BMC Pulm Med. 2015 Dec 24;15:165. doi: 10.1186/s12890-015-0159-z. PMID 26704701
- [Derived] O'Byrne PM, Bleecker ER, Bateman ED, Busse WW, Woodcock A, Forth R, Toler WT, Jacques L, Lotvall J. Once-daily fluticasone furoate alone or combined with vilanterol in persistent asthma. Eur Respir J. 2014 Mar;43(3):773-82. doi: 10.1183/09031936.00064513. Epub 2013 Oct 17. PMID 24136330
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) meeting eligibility criteria at the Screening visit entered a 4-week Run-in Period for completion of Baseline (BL) safety evaluations and to obtain BL measures of asthma status. Par. were then randomized to a 24-week Treatment Period. 1206 par. were screened, 587 were randomized, and 586 received >=1 dose of study treatment.
Groups:
- FF 200 µg OD: Participants received FF 200 microgram (µg) inhalation powder via a Dry Powder Inhaler (DPI) once daily (OD) in the evening plus placebo via the DISKUS/ACCUHALER twice daily (BID), for 24 weeks. Additionally participants were provided with albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
- FF/VI 200/25 µg OD: Participants received Fluticasone Furoate/Vilanterol (FF/VI) 200/25 µg inhalation powder via a DPI OD in the evening plus placebo via the DISKUS/ACCUHALER BID, for 24 weeks. Additionally participants were provided with albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
- FP 500 µg BID: Participants received Fluticasone Propionate (FP) 500 µg inhalation powder via the DISKUS/ACCUHALER BID plus placebo via a DPI OD in the evening, for 24 weeks. Additionally participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
Period: Overall Study
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Started | 194 | 197 | 195
Completed | 146 | 169 | 161
Not Completed | 48 | 28 | 34
Not completed — Adverse Event | 3 | 7 | 2
Not completed — Lack of Efficacy | 21 | 6 | 18
Not completed — Protocol Violation | 5 | 3 | 5
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Physician Decision | 4 | 8 | 1
Not completed — Withdrawal by Subject | 13 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- FF 200 µg OD: Participants received FF 200 µg inhalation powder via a Dry Powder Inhaler DPI OD in the evening plus placebo via the DISKUS/ACCUHALER BID, for 24 weeks. Additionally participants were provided with albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg inhalation powder via a DPI OD in the evening plus placebo via the DISKUS/ACCUHALER BID, for 24 weeks. Additionally participants were provided with albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
- FP 500 µg BID: Participants received FP 500 µg inhalation powder via the DISKUS/ACCUHALER BID plus placebo via a DPI OD in the evening, for 24 weeks. Additionally participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
- Total: Total of all reporting groups
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID | Total
Number analyzed (Participants) | 194 | 197 | 195 | 586
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized to treatment who received at least one dose of study medication. Randomized participants were assumed to have received study medication unless definitive evidence to the contrary existed.
  Years | 44.6 (14.33) | 46.6 (15.05) | 47.3 (14.06) | 46.2 (14.51)
Gender [Count of Participants; unit: Participants] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized to treatment who received at least one dose of study medication. Randomized participants were assumed to have received study medication unless definitive evidence to the contrary existed.
  Participants
    Female | 113 | 116 | 116 | 345
    Male | 81 | 81 | 79 | 241
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who were randomized to treatment who received at least one dose of study medication. Randomized participants were assumed to have received study medication unless definitive evidence to the contrary existed.
  participants
    African American/African Heritage (HER) | 16 | 16 | 19 | 51
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Japanese/East Asian HER/South East Asian HER | 12 | 15 | 13 | 40
    White | 165 | 165 | 162 | 492
    African American/African Heritage and White | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Trough (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 24-week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 measurement taken at the clinic visit while still on treatment. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 was measured electronically by spirometry in the evening at the Baseline (BL) through Week 24 clinic visits. The highest of 3 technically acceptable measurements was recorded. BL was the pre-dose value obtained at Visit 3. Change from BL was calculated as the Week 24 value minus the Baseline value. The analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of BL trough FEV1, country, sex, age, and treatment group.The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-BL on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of the study medication. Only those participants with non-missing covariates and a post-Baseline FEV1 measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 186 | 187 | 190
Liters | 0.201 (0.0303) | 0.394 (0.0302) | 0.183 (0.0300)
Statistical Analysis 1: Comparison: FF 200 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 0.193, 95% CI 2-sided [0.108 to 0.277]
Statistical Analysis 2: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 0.210, 95% CI 2-sided [0.127 to 0.294]
Statistical Analysis 3: Comparison: FF 200 µg OD vs FP 500 µg BID; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the confidence interval (CI: 0.025, 1-sided significance level) for the mean difference in change from Baseline in clinic visit trough FEV1 of FF 200 µg OD versus FP 500 µg BID was greater than -125 milliliters; Median Difference (Final Values) = 0.018, 95% CI 2-sided [-0.066 to 0.102]

2. Primary Outcome: Change From Baseline in Weighted Mean Serial FEV1 Over 0-24 Hours Post-dose at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at the Baseline and Week 24 clinic visits. Weighted mean was calculated using the 24-hour serial FEV1 measurements that included the pre-dose assessment (within 5 minutes prior to dosing) and the post-dose assessments after 5, 15, and 30 minutes and 1, 2, 3, 4, 5, 12, 16, 20, 23, and 24 hours. At each time point, the highest of 3 technically acceptable measurements was recorded. Baseline was the value obtained at Visit 3. Change from Baseline was calculated as the average Week 24 FEV1 value minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Weighted mean serial FEV1 was calculated in the subset of participants for whom serial FEV1 at Week 24 was performed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 83 | 89 | 86
Liters | 0.328 (0.0493) | 0.464 (0.0470) | 0.258 (0.0483)
Statistical Analysis 1: Comparison: FF 200 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p = 0.048, ANCOVA; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [0.001 to 0.270]
Statistical Analysis 2: Comparison: FF/VI 200/25 µg OD vs FP 500 µg BID; Test type: Superiority or Other; p = 0.003, ANCOVA; Median Difference (Final Values) = 0.206, 95% CI 2-sided [0.073 to 0.339]

3. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free and Symptom-free 24-hour Periods at the End of the 24-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). Similarly, asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication/symptoms was considered to be rescue free/symptom free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of periods
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 193 | 197 | 194
Percentage of periods
  Rescue-free 24-hour periods | 26.6 (2.45) | 38.2 (2.42) | 31.9 (2.45)
  Symptom-free 24-hour periods | 21.0 (2.32) | 29.3 (2.29) | 24.5 (2.31)

4. Secondary Outcome: Change From Baseline in the Total Asthma Quality of Life Questionnaire (AQLQ) (+12) Score at Week 12 and Week 24/Early Withdrawal
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire used to evaluate the impact of asthma treatments on the quality of life of asthma sufferers. The AQLQ for 12 years and older (AQLQ [+12]) is a modified version of the AQLQ for use in asthma patients between the age of 12 and 70. The AQLQ contains 32 items in 4 domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). For the 32 items on the questionnaire, the response format consists of a seven-point scale, where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment." The AQLQ total score is defined as the average of the scores from all 32 questions; thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment"). Baseline was the total score obtained at Visit 3. Change from Baseline was calculated as the total score at Weeks 12 and 24 minus the total score at Baseline.
Time Frame: Baseline, Week 12, and Week 24/Early Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
Scores on a scale
  Week 12, n=154, 180, 163 | 0.66 (0.061) | 0.74 (0.056) | 0.74 (0.059)
  Week 24, n=140, 167, 156 | 0.88 (0.071) | 0.93 (0.065) | 0.90 (0.068)

5. Other Pre Specified Outcome: Clinic Visit 12-hour Post-dose FEV1at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. 12-hour post-dose FEV1 measurements were taken electronically by spirometry at the Week 24 clinic visit. The highest of 3 technically acceptable measurements was recorded.
Time Frame: Week 24
Population: ITT Population. 12-hour post-dose FEV1 was analyzed in the subset of participants for whom serial FEV1 at Week 24 was performed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 82 | 93 | 87
Liters | 2.611 (0.8437) | 2.683 (0.9758) | 2.262 (0.7786)

6. Other Pre Specified Outcome: Change From Baseline in Weighted Mean Serial FEV1 Over 0 to 4 Hours Post-dose at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at Baseline. Weighted mean was calculated using the 4-hour serial FEV1 measurements that included the pre-dose assessment (within 5 minutes prior to dosing) and post-dose assessments after 5, 15, and 30 minutes and 1, 2, 3, and 4 hours. At each time point, the highest of 3 technically acceptable measurements was recorded. Baseline was the value obtained at Visit 3. Change from Baseline was calculated as the average Week 24 FEV1 value minus the Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 83 | 89 | 86
Liters | 0.363 (0.4690) | 0.492 (0.5671) | 0.256 (0.4679)

7. Other Pre Specified Outcome: Mean Change From Baseline in Daily Morning Trough (AM) and Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the First 12 Weeks and 24 Weeks of the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Trough PEF is the PEF measured approximately 24 hours after the last administration of study drug. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily trough AM/PM PEF over 12 weeks and 24 weeks of the 24-week Treatment Period (at Weeks 12 and 24) minus the Baseline value.
Time Frame: From Baseline up to Week 12 and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
Liters/minute (L/min)
  AM PEF, Week 1 to 12, n=193, 197, 195 | 15.1 (2.82) | 48.1 (2.78) | 17.1 (2.80)
  AM PEF, Week 1 to 24, n=193, 197, 195 | 18.2 (2.97) | 51.8 (2.94) | 18.8 (2.95)
  PM PEF, Week 1 to 12, 192, 197, 194 | 7.5 (2.80) | 36.6 (2.75) | 12.6 (2.78)
  PM PEF, Week 1 to 24, 192, 197, 194 | 9.1 (2.98) | 39.8 (2.93) | 13.6 (2.96)

8. Other Pre Specified Outcome: The Number of Participants Who Withdrew Due to Lack of Efficacy During the 24-week Treatment Period
Description: The number of participants whose primary reason for withdrawal was lack of efficacy was analyzed.
Time Frame: From the first dose of the study medication up to Week 24/Early Withdrawal
Population: ITT Population
Measure: Number; unit: participants
Groups:
- FF 200 µg OD Arm: Participants received FF 200 µg inhalation powder via a Dry Powder Inhaler DPI OD in the evening plus placebo via the DISKUS/ACCUHALER BID, for 24 weeks. Additionally participants were provided with albuterol/salbutamol inhalation aerosol to be used as rescue medication as needed.
Arm/Group | FF 200 µg OD Arm | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
participants | 21 | 6 | 18

9. Other Pre Specified Outcome: Change From Baseline in the Asthma Control Test (ACT) Scores at Week 12 and Week 24
Description: The ACT is a 5-item questionnaire developed as a measure of the participant's asthma control. Questions are designed to be self-completed by the participant and include the following: In the past 4 weeks, "How much of the time did your asthma keep you from getting as much done at work, school or at home?", "How often have you had shortness of breath?", "How often did your asthma symptoms wake you up at night or earlier than usual in the morning?", "How often have you used your rescue inhaler or nebulizer medication (such as albuterol)?" and "How would you rate your asthma control"? The ACT total score is defined as the sum of the scores from all 5 questions, provided all questions have been answered; thus, the total score ranges from 5 (poor control of asthma) to 25 (complete control of asthma). A score of 20 or higher indicates well-controlled asthma. Change from Baseline was calculated as the total score at Week 12 and Week 24/Early Withdrawal minus the total score at Baseline.
Time Frame: Baseline, Week 12, and Week 24/Early Withdrawal
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
Scores on a scale
  Week 12, n=164, 183, 169 | 3.9 (0.29) | 4.8 (0.27) | 3.9 (0.28)
  Week 24, n=147, 170, 162 | 5.2 (0.30) | 5.5 (0.28) | 4.7 (0.29)

10. Other Pre Specified Outcome: Number of Participants With the Indicated Global Assessment of Change Questionnaire Responses at Weeks 4, 12, and 24
Description: At the end of Week 4, Week 8, and Week 24/Early Withdrawal, the Global Assessment of Change Questionnaire that assesses changes in asthma symptoms (AS) and rescue medication use (RMU) was completed by the participants. The number of participants who chose the following answers to the questionnaire were determined: much better, somewhat better, a little better, the same, a little worse, somewhat worse, much worse (to assess the changes in asthma symptoms); much less often, somewhat less often, a little less often, the same, a little more often, somewhat more often, much more often (to assess the changes in the frequency of rescue medication use).
Time Frame: Week 4, Week 12, and Week 24/Early Withdrawal
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
participants
  Week 4, AS: Much better, n=174, 191, 180 | 37 | 58 | 35
  Week 4, AS: Somewhat better, n=174, 191, 180 | 47 | 65 | 49
  Week 4, AS: A little better, n=174, 191, 180 | 43 | 34 | 40
  Week 4, AS: The same, n=174, 191, 180 | 35 | 25 | 44
  Week 4, AS: A little worse, n=174, 191, 180 | 8 | 7 | 6
  Week 4, AS: Somewhat worse, n=174, 191, 180 | 2 | 2 | 3
  Week 4, AS: Much worse, n=174, 191, 180 | 2 | 0 | 3
  Week 4, RMU: Much less often, n=174, 191, 180 | 49 | 71 | 42
  Week 4, RMU: Somewhat less often, n=174, 191, 180 | 29 | 48 | 41
  Week 4, RMU: A little less often, n=174, 191, 180 | 42 | 38 | 45
  Week 4, RMU: The same, n=174, 191, 180 | 34 | 27 | 37
  Week 4, RMU: A little more often, n=174, 191, 180 | 14 | 4 | 9
  Week 4, RMU: Somewhat more often, n=174, 191, 180 | 5 | 2 | 3
  Week 4, RMU: Much more often, n=174, 191, 180 | 1 | 1 | 3
  Week 12, AS: Much better, n=162, 183, 165 | 60 | 78 | 54
  Week 12, AS: Somewhat better, n=162, 183, 165 | 43 | 51 | 52
  Week 12, AS: A little better, n=162, 183, 165 | 27 | 33 | 34
  Week 12, AS: The same, n=162, 183, 165 | 23 | 15 | 16
  Week 12, AS: A little worse, n=162, 183, 165 | 8 | 5 | 6
  Week 12, AS: Somewhat worse, n=162, 183, 165 | 0 | 1 | 3
  Week 12, AS: Much worse, n=162, 183, 165 | 1 | 0 | 0
  Week 12, RMU: Much less often, n=162, 183, 164 | 66 | 90 | 59
  Week 12, RMU: Somewhat less often, n=162, 183, 164 | 31 | 36 | 37
  Week 12, RMU: A little less often, n=162, 183, 164 | 28 | 24 | 40
  Week 12, RMU: The same, n=162, 183, 164 | 26 | 24 | 20
  Week 12, RMU: A little more often, n=162, 183, 164 | 7 | 8 | 6
  Week 12, RMU: Somewhat more often, n=162, 183, 164 | 2 | 0 | 1
  Week 12, RMU: Much more often, n=162, 183, 164 | 2 | 1 | 1
  Week 24, AS: Much better, n=146, 168, 162 | 64 | 89 | 62
  Week 24, AS: Somewhat better, n=146, 168, 162 | 43 | 37 | 52
  Week 24, AS: A little better, n=146, 168, 162 | 22 | 23 | 17
  Week 24, AS: The same, n=146, 168, 162 | 11 | 14 | 23
  Week 24, AS: A little worse, n=146, 168, 162 | 3 | 4 | 4
  Week 24, AS: Somewhat worse, n=146, 168, 162 | 2 | 1 | 2
  Week 24, AS: Much worse, n=146, 168, 162 | 1 | 0 | 2
  Week 24, RMU: Much less often, n=146, 168, 162 | 68 | 87 | 69
  Week 24, RMU: Somewhat less often, n=150, 187, 18 | 33 | 38 | 37
  Week 24, RMU: A little less often, n=150, 187, 18 | 29 | 22 | 26
  Week 24, RMU: The same, n=146, 168, 162 | 12 | 16 | 19
  Week 24, RMU: A little more often, n= 142, 168, 16 | 1 | 3 | 8
  Week 24, RMU: Somewhat more often, n=146, 168, 162 | 3 | 1 | 1
  Week 24, RMU: Much more often, n=146, 168, 162 | 0 | 1 | 2

11. Other Pre Specified Outcome: Number of the Indicated Unscheduled Asthma-related Healthcare Visits During the Treatment Period
Description: All unscheduled asthma-related visits to a physician's office, visits to urgent care, visits to the emergency department, and hospitalizations (ICU=intensive care unit; GW=general ward) associated with severe asthma exacerbations or other asthma-related healthcare issues were recorded.
Time Frame: From Baseline up to Week 24/Withdrawal Visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Number analyzed (Participants) | 194 | 197 | 195
Number of visits
  Number of Home Visits (Day) | 0.0 (0.07) | 0.0 (0.00) | 0.0 (0.00)
  Number of Home Visits (Night) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Physician Office/Practice Visits | 0.0 (0.10) | 0.0 (0.00) | 0.1 (0.45)
  Number of Urgent Care/Outpatient Clinic Visits | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Emergency Room Visits | 0.0 (0.07) | 0.0 (0.00) | 0.0 (0.00)
  Number of Inpatient Hospitalization Days (ICU) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Number of Inpatient Hospitalization (GW) Days | 0.0 (0.29) | 0.0 (0.00) | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the the treatment period (up to Week 24).
Description: An on-therapy AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | FF 200 µg OD | FF/VI 200/25 µg OD | FP 500 µg BID
Serious Adverse Events (participants affected / at risk) | 1/194 | 6/197 | 2/195
Other Adverse Events (participants affected / at risk) | 66/194 | 62/197 | 73/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 200 µg OD (N=194) | FF/VI 200/25 µg OD (N=197) | FP 500 µg BID (N=195)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 200 µg OD (N=194) | FF/VI 200/25 µg OD (N=197) | FP 500 µg BID (N=195)
Nasopharyngitis (Infections and infestations) | 27 | 25 | 39
Respiratory tract infection viral (Infections and infestations) | 7 | 7 | 7
Influenza (Infections and infestations) | 8 | 5 | 7
Bronchitis (Infections and infestations) | 6 | 7 | 6
Sinusitis (Infections and infestations) | 7 | 3 | 4
Pharyngitis (Infections and infestations) | 2 | 4 | 6
Rhinitis (Infections and infestations) | 2 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 4
Headache (Nervous system disorders) | 13 | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.